CLINICAL TRIAL: NCT07347938
Title: A Multicenter, Prospective, Non-Randomized, Open-Label, Active-Controlled Phase 4 Study to Evaluate the Effectiveness and Safety of Siltartoxatug Injection for Tetanus Prophylaxis Following Injury
Brief Title: A Phase 4 Study to Evaluate the Effectiveness and Safety of Siltartoxatug Injection for Tetanus Prophylaxis Following Injury
Status: Not yet recruiting | Type: Observational
Sponsor: Zhuhai Trinomab Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: TNM002-401
Record Dates: First submitted 2025-12-25; First posted 2026-01-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2025-12

CONDITIONS: Tetanus
MeSH Terms: conditions — Tetanus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Siltartoxatug Injection: Participants receiving siltartoxatug for tetanus prophylaxis and meeting eligibility criteria will be assigned to the siltartoxatug group (n=4,000).
  Interventions: Drug: Siltartoxatug Injection
- HTIG, TAT, or F(ab')₂: Participants receiving other passive immunizing agents (HTIG, TAT, or F(ab')₂) for tetanus prophylaxis and meeting eligibility criteria will be assigned to the control group (n=2,000), comprising approximately 1,000 HTIG recipients and 1,000 TAT/F(ab')₂ recipients
  Interventions: Drug: HTIG/TAT/F(ab')₂

INTERVENTIONS:
Drug: Siltartoxatug Injection — Dosage form: Injectable solution Strength: 10 mg / 0.5 mL per vial Route and regimen: Single intramuscular injection in the gluteal muscle at a dose of 10 mg
  Groups: Siltartoxatug Injection
Drug: HTIG/TAT/F(ab')₂ — Dosage form, strength, and administration: As specified in the respective product's approved labeling (package insert). All use will follow routine clinical practice per local guidelines.
  Groups: HTIG, TAT, or F(ab')₂

SUMMARY:
Study sites were selected from hospitals across diverse regions of China. Approximately 6,000 participants who require passive immunization against tetanus due to various injuries (including those with severe wounds or heavily contaminated injuries) will be enrolled. Per clinical practice:

Participants receiving siltartoxatug for tetanus prophylaxis and meeting eligibility criteria will be assigned to the siltartoxatug group (n=4,000); Participants receiving other passive immunizing agents (HTIG, TAT, or F(ab')₂) for tetanus prophylaxis and meeting eligibility criteria will be assigned to the control group (n=2,000), comprising approximately 1,000 HTIG recipients and 1,000 TAT/F(ab')₂ recipients. All clinical management decisions, including concomitant tetanus vaccination, will be made by investigators per standard clinical practice at each center.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged ≥18 years.
* Receiving siltartoxatug for tetanus prophylaxis per its approved labeling, or receiving another passive immunizing agent (human tetanus immunoglobulin [HTIG], tetanus antitoxin [TAT], or equine F(ab')₂ fragment [F(ab')₂]) for tetanus prophylaxis per its labeling.
* Receiving or planned to receive standard wound management.
* Providing written informed consent by the subject or their legally authorized representative.

Exclusion Criteria:

* Life expectancy <3 months.
* Severe cognitive impairment or other condition interfering with the assessment of tetanus development.
* Currently participating in another interventional clinical trial (observational studies are permitted).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults (≥18 years of age) who require passive immunization against tetanus following injury.
Sampling Method: Non-Probability Sample
Enrollment: 6000 (Estimated)
Dates: Start 2026-01-05 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-03-31 (Estimated)

PRIMARY OUTCOMES:
Primary Objective | within 90 days
  Tetanus protection rate (1 - tetanus incidence rate) within 90 days post-dosing

SECONDARY OUTCOMES:
Secondary Objective | within 28 days
  Tetanus protection rate (1 - tetanus incidence rate) within 28 days post-dosing
Secondary Objective | within 90 days
  Incidence rates of adverse events (AEs) and serious adverse events (SAEs)

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Affiliated Hospital Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided